CLINICAL TRIAL: NCT03582683
Title: A Randomized Controlled Trial of a Community-Based Chronic Pain Self-Management Program in West Virginia
Brief Title: A Community-Based Chronic Pain Self-Management Program in West Virginia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West Virginia University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); West Virginia School of Osteopathic Medicine (Other); Mid-Ohio Valley Health Department (Unknown)
Responsible Party: Principal Investigator, Dina L Jones, PT, PhD, Professor, West Virginia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 3U48DP005004-04S1 (NIH)
Record Dates: First submitted 2018-06-14; First posted 2018-07-11 (Actual); Last update posted 2021-04-12 (Actual); Status verified 2021-04

CONDITIONS: Chronic Pain
Keywords: Self-Management Programs; Behavioral Health
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: After a baseline assessment, participants will be randomized to the CPSMP intervention or a 6-month, wait-list control group based on an allocation sequence based on class size, that will be stratified by site and allocated via opaque envelopes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CPSMP Intervention (Experimental): Participants randomly assigned to this arm will, following a baseline assessment, immediately begin attending a 6-week Chronic Pain Self-Management Program (CPSMP) workshop.
  Interventions: Behavioral: Chronic Pain Self-Management Program (CPSMP)
- Wait-list Control Group (Active Comparator): Participants assigned to this arm will wait six months after a baseline assessment and then attend the 6-week Chronic Pain Self-Management Program (CPSMP) workshop.
  Interventions: Behavioral: Chronic Pain Self-Management Program (CPSMP)

INTERVENTIONS:
Behavioral: Chronic Pain Self-Management Program (CPSMP) — Stanford University's Chronic Pain Self-Management Program (CPSMP) was developed by Sandra LeFort in 1996 and based on Stanford's Arthritis Self-Management Program and the Chronic Disease Self-Management Program. The 6-week community-delivered workshop consists of 2.5-hour weekly sessions for people with a primary or secondary diagnosis of Chronic Pain.

SUMMARY:
Chronic pain (CP) affects 1 in 3 US adults and costs up to $635 billion annually in medical costs and lost work productivity. Use of opioid medications for CP has risen in the US, and opioid overdose deaths have quadrupled, yet with no overall change in pain. Although one-third of US adults have CP, there is a lack of affordable, non-pharmacological, evidence-based, community-delivered interventions for people with CP.

One program, the Chronic Pain Self-Management Program (CPSMP), provides short-term improvements in pain but its long-term effects have not been evaluated. This study will examine the long-term effects of CPSMP in the medically underserved state of West Virginia (WV). The objectives of this community-engaged, randomized, wait-list controlled study are to: 1) determine the short- (26 weeks) and long-term (52 weeks) effectiveness of the 6-week CPSMP in adults with CP in WV; 2) evaluate the Reach (number of participants, completers), Effectiveness (outcomes), Adoption (number of sites, leaders, trainings), Implementation (fidelity), and Maintenance (satisfaction, continuation) of CPSMP using the RE-AIM Framework; and 3) disseminate the results to key stakeholders including evidence-based organizations, public health practitioners/researchers, and healthcare providers.

The study will enroll 240 participants in 24 workshops at 12 community-based sites in 2 counties in WV, Greenbrier (rural) and Wood (urban). Participants will attend free, 2.5-hour weekly sessions for 6 weeks. Self-reported, performance-based, and physiological data will be collected at baseline and 26, and 52 weeks after the start of the intervention. The primary outcomes are pain (severity, quality, interference, medication use), mental health (mood, anxiety, catastrophizing), function (self-efficacy, coping, health-related quality of life, sleep, fatigue, communication, physical activity), healthcare utilization, missed work days, and gait speed.

DETAILED DESCRIPTION:
Chronic pain (CP) affects 1 in 3 US adults and costs up to $635 billion annually in medical costs and lost work productivity. The impact of CP is worse in people with both CP and comorbid chronic diseases such as arthritis, diabetes, and heart disease. Use of opioid medications for CP has risen in the US, and opioid overdose deaths have quadrupled, yet with no overall change in pain. Although one-third of US adults have CP, there is a lack of affordable, non-pharmacological, evidence-based, community-delivered interventions for people with CP. Thus, there is a vital need to rigorously test more interventions that can be brought to scale and widely disseminated in the US.

One program, the Chronic Pain Self-Management Program (CPSMP), provides short-term improvements in pain but its long-term effects have not been evaluated. This study will examine the long-term effects of CPSMP in the medically underserved state of West Virginia (WV). With one of the worst health profiles in the US, WV has the highest rates of arthritis, diabetes, heart disease, and drug overdose deaths, and therefore has a compelling need for the CPSMP. The objectives of this community-engaged, randomized, wait-list controlled study are to: 1) determine the short- (26 weeks) and long-term (52 weeks) effectiveness of the 6-week CPSMP in adults with CP in WV; 2) evaluate the Reach (number of participants, completers), Effectiveness (outcomes), Adoption (number of sites, leaders, trainings), Implementation (fidelity), and Maintenance (satisfaction, continuation) of CPSMP using the RE-AIM Framework; and 3) disseminate the results to key stakeholders including evidence-based organizations, public health practitioners/researchers, and healthcare providers.

The study will enroll 240 participants in 24 workshops at 12 community-based sites in 2 counties in WV, Greenbrier (rural) and Wood (urban). Participants will attend free, 2.5-hour weekly sessions for 6 weeks. Two trained leaders will facilitate group discussions on managing pain, emotions, depression, fatigue, and sleep; proper exercise, nutrition, and medication use; weight management; strategies for effective communication with healthcare professionals; evaluating treatments; and pacing/planning. Self-reported, performance-based, and physiological data will be collected at baseline and 26, and 52 weeks after the start of the intervention. The primary outcomes are pain (severity, quality, interference, medication use), mental health (mood, anxiety, catastrophizing), function (self-efficacy, coping, health-related quality of life, sleep, fatigue, communication, physical activity), healthcare utilization, missed work days, and gait speed.

ELIGIBILITY:
Inclusion Criteria:

* Adults over age 18
* Have chronic pain (pain on most days or everyday) for the past 3 months or more
* Able to attend 1 CPSMP workshop a week over 6 weeks
* Able to attend 3-4 testing sessions for data collection (testing sessions are scheduled before the workshops begin and then six months, one year and, for those assigned to the control group, one and a half years after the start of the study)

Exclusion Criteria:

* Chronic pain caused by current cancer diagnosis or an open wound
* Lack reliable transportation
* Having surgery for the painful area in the next year
* Not community-dwelling (i.e., living in a nursing home, assisted living or personal care home, mental hospital, or correctional facility)
* Not willing to be randomized to either start CPSMP workshop now or in six months
* Participation in another self-management program (e.g., Diabetes Self-Management Program) in the past 12 months
* Unable to speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2018-06-18 (Actual); Primary Completion 2021-04-09 (Actual); Study Completion 2021-04-09 (Actual)

PRIMARY OUTCOMES:
Pain severity | Change between baseline and 52 weeks
  Using Stanford's 0-10 Pain Visual Numeric Scale participants will rate their pain in the past 2 weeks on an 11-item scale ranging from 0 (no pain) to 10 (severe pain).
Defense and Veterans Pain Rating Scale | Change between baseline and 52 weeks
  Using the Defense and Veterans Pain Rating Scale will rate their pain in the past 2 weeks on an 11-item scale ranging from 0 (no pain) to 10 (severe pain).

SECONDARY OUTCOMES:
Pain interference with sleep | Data will be collected at baseline, 26 weeks after the start of the study and 52 weeks after the study start.
  Defense and Veterans Pain Rating Scale Supplemental Question (revised from 24 hours to past 2 weeks)
Pain frequency | Data will be collected at baseline, 26 weeks after the start of the study and 52 weeks after the study start.
  2016 NHIS (past 3 months)
Perceived disability | Data will be collected at baseline, 26 weeks after the start of the study and 52 weeks after the study start.
  Pain Disability Index
Pain avoidance | Data will be collected at baseline, 26 weeks after the start of the study and 52 weeks after the study start.
  Tampa Scale of Kinesiophobia. A total score is calculated that ranges from 17 (low degree of kinesiophobia) to 68 (a high degree of kinesiophobia)
Opioid misuse | Data will be collected at baseline, 26 weeks after the start of the study and 52 weeks after the study start.
  Screener and Opioid Assessment for Patients with Pain (SOAPP) v1.0-SF
Medication Usage | Data will be collected at baseline, 26 weeks after the start of the study and 52 weeks after the study start.
  Morphine milligram equivalents (MME) per day of current prescription or over-the-counter medications for pain, depression, anxiety, mood, or sleep (also usage of stimulants and muscle relaxers)
Mood | Data will be collected at baseline, 26 weeks after the start of the study and 52 weeks after the study start.
  Stanford Personal Health Questionnaire-Depression (PHQ-8)
Anxiety | Data will be collected at baseline, 26 weeks after the start of the study and 52 weeks after the study start.
  Generalized Anxiety Disorder-7 (GAD-7)
Catastrophizing | Data will be collected at baseline, 26 weeks after the start of the study and 52 weeks after the study start.
  Pain Catastrophizing Scale. The total score ranges from 0 (low catastrophizing) to 52 (high catastrophizing). There are 3 subscales (rumination, magnification, and helplessness)
Mindfulness | Data will be collected at baseline, 26 weeks after the start of the study and 52 weeks after the study start.
  5 Facet Mindfulness Questionnaire Short Form
Pain Self-Efficacy | Data will be collected at baseline, 26 weeks after the start of the study and 52 weeks after the study start.
  Pain Self-Efficacy Scale. The total score ranges from 0 (low self-efficacy) to 60 (high self-efficacy)
Coping | Data will be collected at baseline, 26 weeks after the start of the study and 52 weeks after the study start.
  Coping Strategies Questionnaire-Revised
Activation | Data will be collected at baseline, 26 weeks after the start of the study and 52 weeks after the study start.
  Patient Activation Measure
General Health Status | Data will be collected at baseline, 26 weeks after the start of the study and 52 weeks after the study start.
  2016 BRFSS question
Vitality | Data will be collected at baseline, 26 weeks after the start of the study and 52 weeks after the study start.
  SF-36 v1
Minutes of Physical Activity | Data will be collected at baseline, 26 weeks after the start of the study and 52 weeks after the study start.
  2016 NHIS questions
Healthcare Utilization | Monthly for up to 12 months
  Emergency room visits and doctor/clinic visits
Work | Monthly for up to 12 months
  Number of days missed work and number of days in bed more than half of the day
Gait speed | Data will be collected at baseline, 26 weeks after the start of the study and 52 weeks after the study start.
  5- or 10-meter gait speed test

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - West Virginia School of Osteopathic Medicine, Lewisburg, West Virginia
  - Mid-Ohio Valley Health Department, Parkersburg, West Virginia